CLINICAL TRIAL: NCT01910519
Title: Systems Biology of Influenza A (H5N1) Virus Monovalent Vaccine With and Without AS03 Adjuvant (HIPC: VAX-010)
Brief Title: Systems Biology of Influenza A (H5N1) Virus Monovalent Vaccine With and Without Adjuvant System 03 (AS03)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DAIT HIPC: VAX-010; 1U19AI090023-01 (NIH)
Record Dates: First submitted 2013-07-23; First posted 2013-07-29 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Influenza A Virus, H5N1 Subtype
Keywords: influenza A (H5N1) virus; H5N1 influenza; influenza A/H5/N1; monovalent H5N1 influenza vaccine; systems biology; AS03 adjuvant; unadjuvanted
MeSH Terms: conditions — Influenza in Birds; Virus Diseases | interventions — AS03 adjuvant; Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- H5N1 vaccine plus AS03 adjuvant (Experimental): H5N1 vaccine plus AS03 adjuvant: Influenza A Vaccine with AS03 adjuvant
  Participants receive 2 intramuscular doses of Influenza A (H5N1) Virus Monovalent Vaccine with AS03 adjuvant given 21 days apart (i.e., Administer day 1, booster at Day 21).
  Interventions: Biological: H5N1 vaccine plus AS03 adjuvant
- H5N1 vaccine without adjuvant (Experimental): H5N1 vaccine without adjuvant: Influenza A Vaccine without AS03 adjuvant
  Participants receive 2 intramuscular doses of Influenza A (H5N1) Virus Monovalent Vaccine without AS03 adjuvant given 21 days apart (i.e., Administer day 1, booster at Day 21).
  Interventions: Biological: H5N1 vaccine without adjuvant

INTERVENTIONS:
Biological: H5N1 vaccine plus AS03 adjuvant — Administered vaccine: [GlaxoSmithKline] Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted.
  Participants receive 2 intramuscular doses of Influenza A (H5N1) Virus with AS03 adjuvant, administered 21 (+/- 3) days apart.
  Other Names: Q-Pan H5N1; adjuvanted Q-Pan H5N1
  Arms: H5N1 vaccine plus AS03 adjuvant
Biological: H5N1 vaccine without adjuvant — Administered vaccine: [GlaxoSmithKline] Influenza A (H5N1) Virus Monovalent Vaccine without AS03 adjuvant.
  Participants receive 2 intramuscular doses of Influenza A (H5N1) Virus without adjuvant, administered 21 (+/- 3) days apart.
  Other Names: unadjuvanted H5N1 vaccine
  Arms: H5N1 vaccine without adjuvant

SUMMARY:
This study will compare the different immune responses to Influenza A (H5N1) Virus Monovalent Vaccine with and without the AS03 adjuvant. The Influenza A (H5N1) Virus Monovalent Vaccine with AS03 adjuvant vaccine is approved for use for adults to protect against flu caused by the A/H5N1 "bird flu" virus in Europe but none of the vaccines to be used in the study are approved for use in the United States. The results of this study will help researchers learn about better ways to vaccinate people against the H5N1 flu.

DETAILED DESCRIPTION:
The influenza virus (a germ) causes influenza or "flu." The flu is an infection of the breathing tubes and the lungs. In recent years, flu viruses that at first only infected birds have begun to infect humans. One of these strains is called avian influenza (A/H5N1 subtype) or "bird flu". Although no human cases of bird flu have been diagnosed in the United States, this strain has caused severe illness and death in several hundred people since late 2003. .

Vaccination is the most effective way of controlling flu and preventing its illness and complications. Vaccines help prevent illness by causing the body to make antibodies that fight infection. One way to improve the effectiveness of a vaccine is to include a substance that can stimulate the immune system to make more antibodies. This type of substance is called an adjuvant; one type of adjuvant is called AS03 (Adjuvant System 03).

ELIGIBILITY:
Inclusion Criteria:

* Individuals in good health (as determined by vital signs, medical history, physical examination and laboratory tests);
* Able to understand and give informed consent;
* Women of childbearing potential must agree to practice adequate contraception 1 month prior to study entry and until day 100 of the study.

Exclusion Criteria:

* Personal or family history of sleeping disorders including any of the following: Narcolepsy with or without cataplexy; Idiopathic Hypersomnia or excessive daytime sleepiness of unknown origin; Sleep paralysis; Sleep related hallucinations (hypnagogic or hypnopompic hallucinations);
* Human leukocyte antigen (HLA)-DQB1*06:02 positivity (or DQB1*06 positivity if high resolution HLA testing cannot be performed);
* An abnormal erythrocyte sedimentation rate at baseline;
* Receipt of blood products 3 months prior to study entry and until day 100 of the study;
* Volunteers who donated blood 56 days before screening and have plans to donate on or before day 100 of the study;
* Hemoglobin value of less than 12 mg/dL for females and less than 13 mg/dL for males;
* A positive result in the Narcolepsy Mini Screen questionnaire;
* A score of ≥11 on the Epworth sleepiness scale questionnaire;
* Receipt of any experimental agents within 6 weeks prior to first vaccination and until the completion of the study;
* Receipt of any licensed live vaccine within 4 weeks or any licensed inactivated vaccine within 2 weeks prior to the first study vaccination or planned receipt of any vaccine within 42 days after study entry;
* Receipt of a H5 vaccine or AS03-adjuvanted vaccine at any time in the past prior to current study or have a history of A/H5N1 infection;
* Influenza-like illness (ILI) or documented influenza infection during the 2013-2014 influenza season. [Not excluded from the study, volunteers with prior upper respiratory infections other than ILI];
* Chronic medical problems including (but not limited to) insulin dependent diabetes, severe heart disease, severe lung disease, severe liver disease, severe kidney disease, autoimmune disease, severe gastrointestinal disease;
* Alcohol or drug abuse and psychiatric conditions that in the opinion of the investigator would preclude compliance with the trial or interpretation of safety or endpoint data;
* Impaired immune function or chronic infections including (but not limited to) HIV, hepatitis B or C; organ transplant; active cancer or any history of hematologic cancer; receipt of chemotherapy, radiation therapy (past 36 months) or any other potentially immunosuppressive therapy [i.e. Systemic steroids at any dose and intra-articular administration of steroids in the past 3 months; (Nasal and topical steroids are allowed)], congenital immunodeficiency, anatomical or functional asplenia;
* Heart rate less than 40 bpm or greater than 100 bpm. Systolic blood pressure is less than 90 mm Hg or equal or greater than 160 mm Hg. Diastolic blood pressure is less than 60 mm Hg or equal or greater than 100 mg Hg;
* Pregnancy or postpartum (less than 1 year after delivery) or breast feeding;
* Severe reactions to prior vaccination with influenza virus vaccines, including anaphylaxis;
* History of Guillain-Barré syndrome;
* A previous sudden life-threatening allergic reaction to any ingredient of Influenza A (H5N1) Virus Monovalent Vaccine with or without AS03 adjuvant or to any of the substances that may be present in trace amounts such as thiomersal, egg residues including ovalbumin as well as residual amounts of sodium deoxycholate detergent, formaldehyde and sucrose;
* Volunteers with any acute illness, including any fever (> 100.4 F [> 38.0 C], regardless of the route) within 3 days prior to study entry;
* Social, occupational, or any other condition that in the opinion of the investigator might interfere with compliance with the study and vaccine evaluation.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Rouphael, MD, Principal Investigator — Hope Clinic, Emory University
Locations (1):
- The Hope Clinic - Emory Vaccine Center, Decatur, Georgia, United States

REFERENCES:
- [Derived] Wimmers F, Donato M, Kuo A, Ashuach T, Gupta S, Li C, Dvorak M, Foecke MH, Chang SE, Hagan T, De Jong SE, Maecker HT, van der Most R, Cheung P, Cortese M, Bosinger SE, Davis M, Rouphael N, Subramaniam S, Yosef N, Utz PJ, Khatri P, Pulendran B. The single-cell epigenomic and transcriptional landscape of immunity to influenza vaccination. Cell. 2021 Jul 22;184(15):3915-3935.e21. doi: 10.1016/j.cell.2021.05.039. Epub 2021 Jun 25. PMID 34174187
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized to receive Influenza A (H5N1) Virus Monovalent Vaccine with or without AS03 adjuvant undergoing scheduled anterior cruciate ligament (ACL) surgery at the Hope Clinic - Emory Vaccine Center in Decatur, Georgia. Participants were enrolled between July 2013 and January 2014.
Pre-assignment Details: Of the 99 screened participants, 50 were enrolled and vaccinated. 2 participants withdrew from the study.
Groups:
- Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant: Participants randomized to receive Influenza A (H5N1) Virus Monovalent Vaccine with AS03 adjuvant
- Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv: Participants randomized to receive Influenza A (H5N1) Virus Monovalent Vaccine without AS03 adjuvant
Period: Overall Study
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant | Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv
Started | 35 | 15
Completed | 31 | 15
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant | Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv | Total
Number analyzed (Participants) | 35 | 15 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 15 | 50
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 8 | 30
  Male | 13 | 7 | 20
Region of Enrollment [Number; unit: participants]
  United States | 35 | 15 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in Traditional Immune Parameters Measurements Using Luminex Assays and Gene Expression Measurement Using Microarray Experiments From Baseline With Influenza A Vaccine With and Without AS03 Adjuvant
Description: To identify innate immune signatures; 1 day post first vaccination
Time Frame: Day 1
Measure: Number; unit: differentially expressed genes (DEGs)
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant | Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv
Number analyzed (Participants) | 35 | 15
differentially expressed genes (DEGs)
  Upregulated | 1434 | 128
  Downregulated | 1768 | 56

2. Primary Outcome: Change in Traditional Immune Parameters Measurements Using Luminex Assays and Gene Expression Measurement Using Microarray Experiments From Baseline With Influenza A Vaccine With and Without AS03 Adjuvant
Description: To identify innate immune signatures; 3 days post first vaccination
Time Frame: Day 3
Measure: Number; unit: differentially expressed genes (DEGs)
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant | Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv
Number analyzed (Participants) | 35 | 15
differentially expressed genes (DEGs)
  Upregulated | 654 | 787
  Downregulated | 445 | 620

3. Primary Outcome: Change in Traditional Immune Parameters Measurements Using Luminex Assays and Gene Expression Measurement Using Microarray Experiments From Baseline With Influenza A Vaccine With and Without AS03 Adjuvant
Description: To identify innate immune signatures; 7 days post first vaccination
Time Frame: Day 7
Measure: Number; unit: differentially expressed genes (DEGs)
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant | Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv
Number analyzed (Participants) | 35 | 15
differentially expressed genes (DEGs)
  Upregulated | 149 | 83
  Downregulated | 232 | 178

4. Primary Outcome: Change in Traditional Immune Parameters Measurements Using Luminex Assays and Gene Expression Measurement Using Microarray Experiments From Baseline With Influenza A Vaccine With and Without AS03 Adjuvant
Description: To identify innate immune signatures; 1 day post second vaccination
Time Frame: Day 22
Measure: Number; unit: differentially expressed genes (DEGs)
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant | Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv
Number analyzed (Participants) | 35 | 15
differentially expressed genes (DEGs)
  Upregulated | 1953 | 81
  Downregulated | 2820 | 99

5. Primary Outcome: Change in Traditional Immune Parameters Measurements Using Luminex Assays and Gene Expression Measurement Using Microarray Experiments From Baseline With Influenza A Vaccine With and Without AS03 Adjuvant
Description: To identify innate immune signatures; 3 days post second vaccination
Time Frame: Day 24
Measure: Number; unit: differentially expressed genes (DEGs)
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant | Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv
Number analyzed (Participants) | 35 | 15
differentially expressed genes (DEGs)
  Upregulated | 839 | 78
  Downregulated | 487 | 172

6. Primary Outcome: Change in Traditional Immune Parameters Measurements Using Luminex Assays and Gene Expression Measurement Using Microarray Experiments From Baseline With Influenza A Vaccine With and Without AS03 Adjuvant
Description: To identify innate immune signatures; 7 days post second vaccination
Time Frame: Day 28
Measure: Number; unit: differentially expressed genes (DEGs)
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant | Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv
Number analyzed (Participants) | 35 | 15
differentially expressed genes (DEGs)
  Upregulated | 63 | 34
  Downregulated | 28 | 52

7. Primary Outcome: Measurement of Hemagglutination Inhibition Assay (HAI) Titers With Influenza A Vaccine With and Without AS03 Adjuvant
Description: To measure selective adaptive immune response; 21 days post first vaccination
Time Frame: Day 21
Measure: Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant | Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv
Number analyzed (Participants) | 35 | 15
IU/ml | 5.561 [4.976 to 6.213] | 5 [5 to 5]

8. Primary Outcome: Measurement of Microneutralization (MN) Titers With Influenza A Vaccine With and Without AS03 Adjuvant
Description: To measure selective adaptive immune response; 21 days post first vaccination
Time Frame: Day 21
Measure: Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant | Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv
Number analyzed (Participants) | 35 | 15
IU/ml | 30.18 [23.08 to 39.47] | 10.44 [9.522 to 11.45]

9. Primary Outcome: Measurement of Hemagglutination Inhibition Assay (HAI) Titers With Influenza A Vaccine With and Without AS03 Adjuvant
Description: To measure selective adaptive immune response; 21 days post second vaccination
Time Frame: Day 42
Measure: Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant | Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv
Number analyzed (Participants) | 35 | 15
IU/ml | 41.3 [26.19 to 65.12] | 5.183 [4.919 to 5.462]

10. Primary Outcome: Measurement of Microneutralization (MN) Titers With Influenza A Vaccine With and Without AS03 Adjuvant
Description: To measure selective adaptive immune response; 21 days post second vaccination
Time Frame: Day 42
Measure: Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant | Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv
Number analyzed (Participants) | 35 | 15
IU/ml | 523.3 [354.5 to 772.5] | 22.78 [13.46 to 38.55]
Statistical Analysis 1: Comparison: Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant vs Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv; Correlation of vaccine-induced blood transcription modules (BTMs) M183-TBA at day 1 with MN titers at day 42; Test type: Other; p = 0.0039, ANOVA
Statistical Analysis 2: Comparison: Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant vs Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv; Correlation of vaccine-induced blood transcription modules (BTMs) M115-cytokines-receptors cluster at day 1 with MN titers at day 42; Test type: Other; p = 0.0368, ANOVA
Statistical Analysis 3: Comparison: Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant vs Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv; Correlation of vaccine-induced blood transcription modules (BTMs) M74-transcriptional targets of glucocorticoid receptor at day 1 with MN titers at day 42; Test type: Other; p = 0.0465, ANOVA
Statistical Analysis 4: Comparison: Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant vs Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv; Correlation of vaccine-induced blood transcription modules (BTMs) M58-B cell development/activation at day 1 with MN titers at day 42; Test type: Other; p = 0.0411, ANOVA
Statistical Analysis 5: Comparison: Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant vs Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv; Correlation of vaccine-induced blood transcription modules (BTMs) M114.0-TBA at day 1 with MN titers at day 42; Test type: Other; p = 0.0067, ANOVA

ADVERSE EVENTS:
Time Frame: Day 0 - Day 7 after 2 intramuscular doses of Influenza A (H5N1) Virus Monovalent Vaccine with or without AS03 adjuvant given 21 days apart.
Description: Local and systemic reactogenicity after receipt of each vaccine
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant | Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/15
Other Adverse Events (participants affected / at risk) | 34/35 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant (N=35) | Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv (N=15)
Missed abortion (unrelated to study vaccine) (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Missed abortion
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Influenza A (H5N1) Virus Monovalent Vaccine With AS03 Adjuvant (N=35) | Influenza A (H5N1) Virus Monovalent Vaccine Without AS03 Adjuv (N=15)
Body ache (General disorders) | 13 (16) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Allergic reaction (Immune system disorders) | 2 (2) | 1 (1)
Upper Respiratory Infections (Infections and infestations) | 2 (2) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (2)
Nausea (General disorders) | 3 (4) | 3 (3)
Malaise (General disorders) | 0 (0) | 1 (1)
Vomiting (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes